CLINICAL TRIAL: NCT07122011
Title: Exploration of Neurophysiological Mechanisms of Exercise-Induced Hypoalgesia With Blood Flow Restriction in Healthy Adults
Brief Title: Neural Contributions to Exercise-Induced Hypoalgesia With Blood Flow Restriction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gran Rosario (Other)
Responsible Party: Principal Investigator, Leonardo Intelangelo, Director, University of Gran Rosario
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Universidad del Gran Rosario
Record Dates: First submitted 2025-08-06; First posted 2025-08-14 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: Blood flow restriction training; Exercise-induced hypoalgesia; Pain modulation; Quantitative sensory testing

STUDY DESIGN:
Intervention Model Description: Single-arm, pre-post experimental study assessing within-subject changes in sensory pain thresholds after a low-load resistance training session with BFR.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group - Low-Intensity Resistance Training with BFR (Experimental): A single session of low-intensity resistance training combined with BFR applied to the proximal thigh of the dominant leg at 60% of total arterial occlusion pressure. Sensory and pain modulation assessments (PPT, CPM, TS, and thermal thresholds) performed immediately before and after the training session.
  Interventions: Other: Low-Intensity Resistance Training with BFR

INTERVENTIONS:
Other: Low-Intensity Resistance Training with BFR — Warm-up: Five minutes of light-intensity cycling on a stationary bike.
  Exercises:
  1. Bilateral half squat (0°-90°)
  2. Single-leg step-down from a 20 cm step
  3. Knee extension (90°-0°) at 30% of one-repetition maximum (1RM)
  4. Single-leg shallow squat (0°-45°)
  Protocol: One set of 30 repetitions (or until volitional fatigue) followed by three sets of 15 repetitions for each exercise.
  Rest periods: One minute between sets and two minutes between exercises.
  BFR Application: Pneumatic cuff (The Occlusion Cuff Pro®) placed proximally on the dominant thigh, inflated to 60% of complete arterial occlusion (determined via Doppler ultrasound). The cuff remains inflated during sets and rest periods, and is deflated after completion of each exercise.

SUMMARY:
This experimental study explores the neurophysiological mechanisms associated with pain modulation following a single session of low-intensity resistance exercise combined with BFR in healthy young adults. The study evaluates changes in sensory thresholds before and after the intervention using validated quantitative sensory testing (QST) methods. These include pressure pain thresholds, conditioned pain modulation, thermal thresholds, and temporal summation. The findings may contribute to a better understanding of the role of the nervous system in exercise-induced hypoalgesia, particularly in response to BFR protocols, with implications for future research in pain and rehabilitation.

DETAILED DESCRIPTION:
Exercise-induced hypoalgesia (EIH) is a physiological response characterized by reduced pain sensitivity following physical activity. Several central and peripheral mechanisms have been proposed to explain EIH, including activation of descending inhibitory pathways and peripheral nociceptor modulation. BFR training involves the application of controlled vascular occlusion during low-load exercise and has shown promising results in enhancing both muscle function and pain modulation.

This is a single-arm, pre-post experimental study involving healthy adults aged 18-35 years. All participants undergo a single session of low-intensity resistance exercise involving the lower limbs, performed under 60% limb occlusion pressure. QST is performed before and immediately after the intervention, including:

Pressure Pain Thresholds (PPT) measured with a digital algometer

Conditioned Pain Modulation (CPM) using cold-water immersion

Thermal thresholds assessed with a computer-controlled thermode

Temporal summation (TS) of pain via repeated pressure stimuli

The aim of this study is to explore the involvement of neurophysiological mechanisms-both central and peripheral-in the pain modulatory response following BFR exercise. This study is conducted at CUADI (Centro Universitario de Asistencia, Docencia e Investigación) in Rosario, Argentina. The results will contribute to basic science knowledge on pain physiology in healthy individuals and may inform future applied research in rehabilitation contexts.

Sample size considerations:

The estimated sample size is approximately 20 participants. This number is based on a preliminary power analysis conducted from pilot data on PPT changes following cold water immersion, which showed a mean difference of 0.77 kgf with a standard deviation of 0.33 kgf. Using G*Power software (v3.1), the calculated sample size for a paired comparison with 95% power and alpha of 0.05 was 16 subjects. To account for potential data loss or dropouts, we plan to include at least 20 individuals. This sample size is considered adequate for a mechanistic, single-arm pre-post design focusing on within-subject changes in pain modulation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic at the time of evaluation.
* Able to provide written informed consent.
* Available to attend a single evaluation and intervention session at the research center.

Exclusion Criteria:

* Bilateral knee symptoms or suspected patellar tendinopathy.
* Increased symptoms with dynamic loading.
* Neurological disorders.
* Inflammatory rheumatic diseases.
* Cardiac diseases.
* Any surgery within the last 3 months.
* Pregnancy.
* Alcohol consumption on the day of participation.
* Hypertension (systolic blood pressure ≥140 mmHg).
* History of deep vein thrombosis.
* History of endothelial dysfunction.
* Peripheral vascular disease.
* Diabetes.
* Active infection.
* Spinal or referred pain.
* Previous experience with blood flow restriction (BFR) training.
* Overweight or obesity.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
CPM | Baseline (before intervention) and immediately after the intervention session.
  Changes in CPM will be assessed by immersing the hand up to the wrist in a cold water bath (0.6-0.8°) with a circulating water pump.The dominant arm for healthy participants will be immersed in the cold-water bath. In general, the conditioning stimulus will be applied for 2 min or maximum tolerance (whichever comes first). A computerized, custom-made visual analog scale will be used to continuously track the response profile to conditional stimuli across participants during the application of CPM. A numeric rating scale ranging from 0 to 100, where 0 represents no perception, 30 represents pain threshold (defined as the time to reach a painful sensation at the predefined stimulation intensity) and 100 represents the tolerance threshold (defined as the sensation of pain when becomes intolerable). Before and immediately after the immersion, PPT measurements will be assessed on medial joint line of the dominant knee and dorsal forearm contralateral to the knee.
PPT | At baseline and immediately after the intervention session.
  Change in PPT will be assessed using a digital algometer (1 cm² round tip) applied perpendicularly to the skin at a rate of 1 kg/s until pain is first perceived. Three measurements will be averaged for each site. Measurement sites include the medial joint line of the dominant knee and the dorsal forearm contralateral to the knee. Each measurement will be performed at 30-second intervals.

SECONDARY OUTCOMES:
Thermal sensitivity thresholds | Immediately before and immediately after the intervention session.
  Changes in heat detection thresholds (HDT, in °C), heat pain thresholds (HPT), and heat pain tolerance thresholds (HTPT) will be assessed by applying heat stimuli to the volar aspect of the non-dominant forearm. Tests will be performed in randomized order. Stimuli will be delivered using a thermode with a 9 cm² contact surface. The baseline temperature will be set at 30 °C, and the skin will be heated at a rate of 1 °C/sec until the first sensation of heat is perceived (HDT), the onset of pain is perceived (HPT), and the pain becomes intolerable (HTPT). The minimum stimulus temperature will be 0 °C, and the maximum will be 50 °C. After reaching the target threshold, the thermode will return to 30 °C at a rate of 5 °C/sec. A 30-second rest interval will be provided before the next measurement. Each test will be repeated three times at each assessment point, with a 30-second interstimulus interval.
TS Score | Immediately before and immediately after the intervention session.
  Changes in TS will be evaluated at the knee and forearm by delivering 10 consecutive pressure pulses at the previously determined PPT intensity, each lasting one second with a one-second interval between pulses. Pain intensity will be rated for the first, fifth, and tenth pulses on a 0-100 numeric rating scale. The TS score will be calculated as the difference between the ratings of the tenth and first pulses.

CONTACTS AND LOCATIONS:
Locations (1):
- University Center for Assistance, Teaching and Research (CUADI), Rosario, Santa Fe Province, Argentina

IPD SHARING:
Plan to Share IPD: Yes
Yes, the statistical analysis plan and informed consent form.
Supporting Information: SAP, ICF
Time Frame: From first date of publication of journal article.
Access Criteria: IPD will be provided upon request.